CLINICAL TRIAL: NCT05120388
Title: Effect of Extra Virgin Olive Oil Addition in the Diet of Women With Gestational Diabetes Mellitus (OLIDIAG)
Acronym: OLIDIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Pharmacological and Botanical Research (Other Government)
Collaborators: Sociedad Argentina de Diabetes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11012021
Record Dates: First submitted 2021-10-14; First posted 2021-11-15 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Gestational Diabetes
Keywords: GDM; Extra Virgin Olive Oil; lipid profile; insulin requirement; postpartum reclassification
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Dietary intervention study: GDM patients receiving a WHO diet with or without addition of extra virgin olive oil
Who Masked: Investigator
Masking Description: Data analysis will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary addition of extra virgin olive oil (Experimental): WHO diet with a daily addition of extra virgin olive oil
  Interventions: Dietary Supplement: Extra Virgin Olive Oil Addition
- No addition of extra virgin Olive Oil (No Intervention): WHO diet

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil Addition — Daily dietary addition of olive oil (three tablespoons)
  Arms: Dietary addition of extra virgin olive oil

SUMMARY:
Gestational diabetes mellitus (GDM) is associated to adverse maternal and neonatal outcomes. The aim of this study is to address whether the addition of extra virgin olive oil to the diet of women with GDM improves maternal triglyceridemia and reduces insulin requirement and diagnosis of diabetes at postnatal reclassification.

DETAILED DESCRIPTION:
This study is a randomized trial in which 1200 pregnant women at GDM diagnosis from 16 health care centers will be recruited and randomized in two parallel arms: 1 World Health Organization (WHO)-diet supplemented with 3 tablespoons of Extra Virgin Olive Oil (Intervention Group, n=600); 2. WHO-diet with no Extra Virgin Olive Oil supplementation (Control Group, n=600). Expected results: the investigators expect that the intervention will contribute to improve maternal lipid profile, reduce insulin requirement and reduce maternal diagnosis of diabetes at postpartum reclassification. Thus, this study is expected to identify maternal beneficial effects of this dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* GDM (diagnosis criteria of the Latin American Society of Diabetes (ALAD) and Argentine Society of Diabetes (SAD): Fasting plasma glucosa > 100 mg/dl, p75 oral glucose tolerance test-2 h plasma glucose > 140 mg/dl)

Exclusion Criteria:

* Multiple pregnancy
* Pregestational diabetes (type 1 or type 2)
* Bariatric surgery
* Infectious diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
maternal triglyceridemia | term pregnancy
  triglycerides in mg/dl
maternal weight gain | change from prepregnancy weight to term pregnancy weight
  gestational maternal weight gain in kg
number of participants with insulin requirement | term pregnancy
  insulin use

SECONDARY OUTCOMES:
number of participants with diabetes at postpartum | six weeks postpartum
  maternal diagnosis of diabetes at postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Patagonica de Medicina Maternofetal y Embarazo de Alto Riesgo, Neuquén, Neuquén Province, Argentina